CLINICAL TRIAL: NCT06142981
Title: Effectiveness of Regenerative Medicine (PRP and PBD-VSEL Stem Cell Therapy) for Parkinson's Disease
Brief Title: PRP and PBD-VSEL Stem Cell Therapy for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Medical University (Other)
Responsible Party: Principal Investigator, Humaira Waseem, Principal Investigator, Fatima Jinnah Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPRM-101
Record Dates: First submitted 2023-11-13; First posted 2023-11-22 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Regenerative Medicine
Keywords: Parkinson's Disease; PRP; Stem cells; Safety
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Patients will receive three PRP sessions, where the patients received intravenous injections at four acupuncture points (stomach 36 and GB 34 on both sides) at the 1st, 2nd, and 3rd month.
  Interventions: Biological: PRP and PBD-VSEL Stem Cell therapy

INTERVENTIONS:
Biological: PRP and PBD-VSEL Stem Cell therapy — The intervention began with the administration of three PRP sessions, where the patients received intravenous injections at four acupuncture points (stomach 36 and GB 34 on both sides) at the 1st, 2nd, and 3rd month.

SUMMARY:
An experimental study will be conducted at Iffat Anwar medical complex conducted to evaluate the effectiveness of PRP and stem Cell therapy in the treatment of PD. After the initial cognitive and laboratory testing, the first infusion appointment will be planned within 2 weeks.

* The treatment began with the administration of three PRP sessions, where the patients received intravenous injections at four acupuncture points (stomach 36 and GB 34 on both sides) at the 1st, 2nd, and 3rd month.
* After three months of treatment, patients were sent back to the neurophysician for evaluation. They will be given a booster dose of PRP during the 1-year follow-up, and then monitored every six months for the next two years.

The primary outcomes of the study will beto see the improvement in The Unified Parkinson's Disease Rating Scale (UPDRS), Hospital Anxiety and Depression Scale (HADS) and self-report Parkinson's Disease Questionnaire-39 (PDQ-39).

DETAILED DESCRIPTION:
Parkinson's disease the second most common neurological disease worldwide is a progressive disorder that affects movement and can cause tremors, stiffness, and difficulty with coordination and balance caused by dopamine deficiency and progressive degeneration of dopaminergic neurons (DAn). Autologous Platelet Rich Plasma (PRP) and Stem cell therapy is new and practical treatment option that aims to decrease neuroinflammation, modulate immune system and stimulate, replace or repair lost or damaged dopamine-producing cells in the brain lost in Parkinson's disease.

Methods:

Total 30 patients aged 30 - 50 years will enrolled in the study. After the initial cognitive and laboratory testing, the patients will be infused PRP in the autologous blood, once a month for 2 months. After three monthly sessions of PRP treatments, peripheral blood derived very small embryonic like (PBD-VSEL) stem cells therapy will be done on the 90th day. All the patients will be sent to neuro physicians for evaluation and improvement after 3 months, 6 months and 12 months.

The primary outcomes of the study will be to see the improvement in The Unified Parkinson's Disease Rating Scale (UPDRS), Hospital Anxiety and Depression Scale (HADS) and self-report Parkinson's Disease Questionnaire-39 (PDQ-39). All the data will be entered and analyzed by SPSS 25.0. Before and after difference outcome variables will compared before and after difference will be observed by paired sample t test. P-value <0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of clinically established PD for at least 1-3 years,
* Both genders aged between 30 to 50 years
* On stable therapy (dopaminergic medication and/or deep brain stimulation parameters)

Exclusion Criteria:

* Gout, congestive heart failure, renal failure
* Uncontrolled atrial fibrillation, stroke, anaphylaxis, blood clotting problem,
* Clinical suspicion or diagnosis of atypical forms of parkinsonism or essential tremor

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
The Unified Parkinson's Disease Rating Scale The Unified Parkinson's Disease Rating Scale | 1 year
  There are four sections of the Unified Parkinson's Disease Rating Scale (UPDRS): four items are used in Part I to assess mentality, behavior, and mood; 13 items are used in Part II to assess activities of daily living; 27 items are used in Part III to measure motor examination; and 11 items are used in Part IV to assess complications of therapy. Each symptom or sign associated with Parkinson's disease is rated on a 5-point Likert scale with scores ranging from 0 to 4.Higher scores indicate more severe impairment. The maximum total UPDRS score of 200 indicates the highest degree of disability caused by Parkinson's disease.
Hospital Anxiety and Depression Scale | 3 to 12 months
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item questionnaire for measuring anxiety and depression. The maximum score for anxiety or depression is 21, with each item having a value between 0 (no impairment) and 3 (significant impairment).
Parkinson's Disease Questionnaire-39 | 1 to 11 months
  The Parkinson's Disease Questionnaire (PDQ-39) assesses the frequency of challenges faced by people with Parkinson's disease in eight areas of daily life, including relationships, social interactions and communication. The PDQ-39 assigns scores on a scale of 0 to 100 for each of the eight dimensions, with higher scores indicating poorer quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: shehzad Anwar, Principal Investigator — University of Lahore
Locations (1):
- gull e Rukh, Lahore, Punjab Province, Pakistan